CLINICAL TRIAL: NCT07256587
Title: Wake Up to Water: Splash Into Morning Energy!
Brief Title: Morning Water Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 37282
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Energy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm longitudinal where participants act as their own control (Experimental): Single Arm longitudinal where participants act as their own control
  Interventions: Other: Drink 24 ounces of water

INTERVENTIONS:
Other: Drink 24 ounces of water — Participants are asked to drink 24 ounces of water first thing upon waking in the morning for 30 days.

SUMMARY:
This study aims to determine the efficacy of morning water consumption on reducing fatigue and boosting daily productivity. Participants will receive personalized feedback on how their morning hydration influences their energy levels, enabling them to make informed decisions on optimizing their daily performance for a more energized life.

ELIGIBILITY:
Inclusion Criteria:

* all individuals over the age of consent

Exclusion Criteria:

* Individuals with Hyponatremia
* Individuals with Kidney Issues
* Individuals with Gastrointestinal Disorders
* Individuals in Occupations with Limited Bathroom Access
* Individuals with Fluid Restrictions
* Individuals Prone to Electrolyte Imbalance

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-23 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
PROMIS Short Form v1.0 - Fatigue 8a | Baseline and 30 days
  PROMIS Short Form v1.0 - Fatigue 8a
Neuro-QOL Item Bank v1.0 -Fatigue - Short Form | Baseline and 30 days
  Neuro-QOL Item Bank v1.0 -Fatigue - Short Form

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is undecided whether this information will be shared yet or not.